CLINICAL TRIAL: NCT06986408
Title: Effect of Earplugs and Eye Masks Used After Orthopedic Surgery on Comfort and Quality of Recovery: A Randomized Controlled Trial
Brief Title: Effect of Earplugs and Eye Masks Used After Orthopedic Surgery on Comfort and Quality of Recovery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Tuba Yılmazer, Assoc. Prof. Dr., Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EarplugsEyeMasks
Record Dates: First submitted 2025-05-14; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Orthopedic Surgery; Nursing Care; Quality of Recovery 40; Comfort
MeSH Terms: interventions — Ear Protective Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Earplugs and Eye Masks (Experimental): The patients in the experimental group will be given the "Informed Consent Form" before surgery and the "Patient Introduction Form" will be applied after permission is obtained. Patients will be given eye masks and earplugs on the nights following surgery and they will be ensured to use them correctly. The "General Comfort Scale" and the "Quality of Recovery Questionnaire (Qor-40)" will be applied 24 and 48 hours after surgery.
  Interventions: Device: Earplugs and Eye Masks
- Standard of care (No Intervention): The patients in the control group will also be given the "Informed Consent Form" before the surgery and the "Patient Introduction Form" will be applied after permission is obtained. The "General Comfort Scale" and the "Quality of Recovery Questionnaire (Qor-40)" will be applied 24 and 48 hours after the surgery. The difference between the groups will be evaluated at the end of the study.

INTERVENTIONS:
Device: Earplugs and Eye Masks — The patients in the experimental group will be given the "Informed Consent Form" before surgery and the "Patient Introduction Form" will be applied after permission is obtained. Patients will be given eye masks and earplugs on the nights following surgery and they will be ensured to use them correctly. The "General Comfort Scale" and the "Quality of Recovery Questionnaire (Qor-40)" will be applied 24 and 48 hours after surgery.
  Arms: Earplugs and Eye Masks

SUMMARY:
This research will be conducted as a randomized controlled trial to determine the effects of earplugs and eye masks used after orthopedic surgery on comfort and quality of recovery. This study is a single-center, parallel-group, open-label, randomized controlled clinical trial. This study will be conducted with 60 patients who underwent orthopedic surgery between June 2025 and October 2025. Participants will be randomized into two equal groups as the intervention group (n=30) and the control group (n=30). The patients in the experimental group will be administered the "Informed Consent Form" and the "Patient Introduction Form" after obtaining permission before surgery. Patients will be given an eye mask and earplugs on the nights following surgery and will be ensured to use them correctly. The "General Comfort Scale" and the "Quality of Recovery Questionnaire (Qor-40)" will be administered 24 and 48 hours after surgery. The patients in the control group will also be administered the "Informed Consent Form" and the "Patient Introduction Form" after obtaining permission before surgery. The "General Comfort Scale" and the "Quality of Recovery Questionnaire (Qor-40)" will be administered 24 and 48 hours after surgery. At the end of the study, the difference between the groups will be evaluated. In the analysis of this study, descriptive statistics, Shapiro-Wilk test, Chi-square test, t-test in independent groups, ANOVA test in repeated measures will be used.

The main questions it aims to answer:

Do earplugs and eye masks used after orthopedic surgery have an effect on comfort level? Do earplugs and eye masks used after orthopedic surgery have an effect on the quality of recovery?

DETAILED DESCRIPTION:
In the postoperative period, patients may experience problems such as pain due to surgery, prolonged fasting, and discomfort caused by foreign equipment (catheter, drain) in their bodies. This situation further exacerbates the existing pain of the patients and reduces their comfort levels. Using more opioids to reduce increased pain negatively affects biological processes such as early mobilization and early nutrition, which are important for the recovery of surgical patients. Therefore, non-pharmacological and non-invasive nursing care practices are needed to increase the comfort levels and quality of recovery of surgical patients. Patients' comfort levels and quality of recovery decrease significantly due to environmental factors such as alarm sounds of devices, high staff turnover, and constantly on lights. When the literature is examined, it is seen that tools and equipment are needed to manage this very important problem. It has been reported that the use of eye masks and earplugs may be better than other interventions in reducing noise and controlling light. The use of eye masks and earplugs is one of the effective and independent nursing interventions. Non-pharmacological tools such as earplugs and eye masks isolate the patient from noise and light. While the effects of using tools and equipment alone or together on the comfort level are discussed in the literature to a limited extent; no study has been found evaluating the effect on the quality of recovery. In the study conducted by Altıntaş et al., it was determined that the comfort levels of the patients increased after the interventions of ergonomic sleep masks, earplugs and eye masks. In some studies, it has been reported that these devices are not comfortable despite their positive effects. While patients may wake up involuntarily when the earplug is removed during sleep, there are also cases where eye masks are not the right size for the patients' head structure and the rope part of the masks is thin and tight, which can disturb the patient. It is important that the use of eye masks and earplugs can be adjusted according to the head and ear structure in terms of patient comfort. For this reason, it is necessary to use ergonomic materials that facilitate patient adaptation, can be adjusted according to the individual, and are reusable in terms of cost effectiveness. While the effects of using earplugs and eye masks on the comfort level of patients are discussed in a limited way in the literature; no study has been found evaluating their effects on the quality of recovery. In addition, no study has been found that determines the effect of earplugs and eye masks used after orthopedic surgery on comfort and healing quality. Based on this point, it was aimed to determine the effect of earplugs and eye masks used after orthopedic surgery on comfort and healing quality.

ELIGIBILITY:
Inclusion Criteria:

* Patients who can speak and understand Turkish,
* At least 18 years old,
* No hearing impairment and not using hearing aids,
* No psychiatric diagnosis and not using psychiatric medication regularly,
* Patients who agree to participate in the study and have given written consent.

Exclusion Criteria:

* Patients who do not agree to participate in the study and for whom written consent was not obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
General Comfort Scale Short Form | just 24 and 48 hours
  The scale describes individual comfort needs and the components of the concept of comfort for nursing as relief, relaxation, and overcoming problems. The highest total score that can be obtained from the scale is 168 points; the lowest total score is 28 points. A low score from the scale indicates a low comfort level.
Quality of Recovery Scale (Qor-40) | just 24 and 48 hours
  This scale is a 40-question survey and includes five sub-dimensions, 'Emotional State, Physical Comfort, Patient Support, Physical Independence and Pain', to evaluate the individual's own condition, pain intensity and physical and emotional conditions. The total survey score varies between 40 and 200. An increase in the total score given to the survey indicates that individuals are doing well at the expected level in the post-surgical period.